CLINICAL TRIAL: NCT02132910
Title: Restorative Exercise for Strength Training and Operational Resilience
Brief Title: Restorative Exercise for Strength Training and Operational Resilience (RESTORE) for Chronic or Recurrent Low Back Pain
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 380491
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

ARMS (2):
- RESTORE Intervention (Experimental): 1. First you will receive an initial assessment of pain, physical function, and behavioral health. You will be asked to take a computer questionnaire, perform some simple physical assessments, and answer questions about yourself, your pain and your current medication use.
  2. For the first four weeks you will receive twice-weekly, individualized, hour-long RESTORE sessions from a specially trained RESTORE instructor.
  3. For the next four weeks, you will receive weekly, individualized, hour-long RESTORE sessions from a RESTORE instructor.
  4. At weeks four and eight, you will repeat the assessment of pain, physical function, and behavioral health. You will be asked to take a computer questionnaire, perform some simple physical assessments, and answer questions about pain and medication use.
  5. At three and six months, you will be contacted by telephone or email to answer questionnaires about pain, physical function, and behavioral health.
  Interventions: Other: RESTORE Intervention
- Control Group 2 (No Intervention): 1. First you will receive an initial assessment of pain, physical function, and behavioral health. You will be asked to take a computer questionnaire, perform so simple physical assessments, and answer questions about yourself, your pain and your current medication use.
  2. You will be contacted once a week for eight weeks by phone or email to answer questions about your pain level.
  3. At weeks four and eight, you will repeat the assessment of pain, physical function and behavioral health. You will be asked to take a computer questionnaire, perform some simple physical assessments, and answer questions about pain and medication use.
  4. At three and six months, you will be contacted by telephone or email to answer questionnaires about pain, physical function, and behavior health.

INTERVENTIONS:
Other: RESTORE Intervention
  Arms: RESTORE Intervention

SUMMARY:
The purpose of the study is to learn about the effect of integrative therapies on chronic or recurrent low back pain.

The intervention called RESTORE (Restorative Exercises for Strength Training and Operational Resilience) is based on a series of gentle stretching and strengthening exercises incorporating breath-work and mindfulness. The study is designed to discover the impact of RESTORE on pain levels, physical function, and behavioral health.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lower back pain with a pain score of 4 or higher on DVPRS for 3 months
* Male or female
* Age 18-68*
* Able to read and understand English
* Understands language, and able to report current pain levels and recall events
* DEERS-Eligible, Military healthcare beneficiary

Exclusion Criteria:

* Provider has advised against mild to moderate exercise
* Patient unable to sit on the floor for two minutes or unable to stand independently
* Complex Regional Pain Syndrome, Fibromyalgia, Chronic Fatigue Syndrome, Auto Immune disease-related pain, other chronic medical conditions (i.e. advanced diabetic neuropathies) that preclude consent
* Patients with severe TBI
* Practiced Yoga within 6 months
* Pre-surgical candidates for back surgery within 3 months
* Back surgery within the past year
* Pregnancy**; females will be asked to self-report
* Undergoing Medical Evaluation Board to determine discharge

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08-07 (Actual); Study Completion 2015-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chester Buckenmaier, MD, Principal Investigator — Defense and Veterans Center for Integrative Pain Management
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Highland KB, Schoomaker A, Rojas W, Suen J, Ahmed A, Zhang Z, Carlin SF, Calilung CE, Kent M, McDonough C, Buckenmaier CC 3rd. Benefits of the Restorative Exercise and Strength Training for Operational Resilience and Excellence Yoga Program for Chronic Low Back Pain in Service Members: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Jan;99(1):91-98. doi: 10.1016/j.apmr.2017.08.473. Epub 2017 Sep 14. PMID 28919191

RESULTS

PARTICIPANT FLOW:
Groups:
- RESTORE Intervention: 1. First you will receive an initial assessment of pain, physical function, and behavioral health. You will be asked to take a computer questionnaire, perform some simple physical assessments, and answer questions about yourself, your pain and your current medication use.
  2. For the first four weeks you will receive twice-weekly, individualized, hour-long RESTORE sessions from a specially trained RESTORE instructor.
  3. For the next four weeks, you will receive weekly, individualized, hour-long RESTORE sessions from a RESTORE instructor.
  4. At weeks four and eight, you will repeat the assessment of pain, physical function, and behavioral health. You will be asked to take a computer questionnaire, perform some simple physical assessments, and answer questions about pain and medication use.
  5. At three and six months, you will be contacted by telephone or email to answer questionnaires about pain, physical function, and behavioral health.
  RESTORE Intervention
Period: Overall Study
Arm/Group | RESTORE Intervention | Control Group 2
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RESTORE Intervention | Control Group 2 | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 65
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 15 | 10 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Participants will choose a pain score using the Defense and Veteran's Pain Rating Scale 2.0
  Rate the severity of your CURRENT pain:
  0 - No Pain
  1. - Hardly notice pain
  2. - Notice pain, does not interfere with activities
  3. - Sometimes distracts me
  4. - Distracts me, can do usual activities
  5. - Interrupts some activities
  6. - Hard to ignore, avoid usual activities
  7. - Focus of attention, prevents doing daily activities
  8. - Awful, hard to do anything
  9. - Can't bear pain, unable to do anything
  10. - As bad as it could be, nothing else matters
  Higher values represent worse outcomes
Time Frame: Baseline, Midtreatment, Posttreatment, 3 month follow-up, 6 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group 2 | RESTORE Intervention
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 4.32 (1.61) | 4.68 (1.51)
  Midtreatment | 3.97 (1.71) | 2.60 (1.83)
  Posttreatment | 3.67 (1.86) | 2.48 (2.34)
  3 month follow up | 3.35 (1.79) | 2.75 (2.43)
  6 month follow up | 2.86 (2.01) | 2.79 (2.34)

2. Secondary Outcome: Disability
Description: The Roland Morris Disability Questionnaire is reliable at measuring level of disability and is sensitive to change over time for groups of patients with lower back pain.
  Scale: 0-24 (24 total statements)
  -Greater levels of disability are reflected by higher numbers on a 24-point scale See link for complete statements: https://www.worksafe.qld.gov.au/__data/assets/pdf_file/0009/76851/roland-morris-low-back-pain-and-disability-questionnaire-rmq1.pdf
Time Frame: Baseline, Midtreatment, Posttreatment, 3 month follow up, 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group 2 | RESTORE Intervention
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 8.68 (4.82) | 9.21 (4.91)
  Midtreatment | 8.03 (5.46) | 5.90 (4.52)
  Posttreatment | 6.70 (4.59) | 4.41 (4.67)
  3 month follow up | 7.04 (4.55) | 4.43 (4.62)
  6 month follow up | 6.52 (5.33) | 3.25 (3.15)

3. Other Pre Specified Outcome: Physical Functioning
Description: Physical functioning was assessed using the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Physical Functioning subscale (0-100) Total scores are transformed to standardized t scores (mean=50; SD=10). Higher scores indicate higher physical functioning.
Time Frame: Baseline, Midtreatment, Posttreatment, 3 month follow up, 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group 2 | RESTORE Intervention
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 42.03 (5.29) | 40.67 (3.71)
  Midtreatment | 42.71 (6.16) | 45.79 (7.10)
  Posttreatment | 42.72 (5.55) | 47.44 (7.44)
  3 month follow up | 43.38 (4.82) | 47.34 (7.43)
  6 month follow up | 44.06 (6.66) | 47.05 (8.00)

4. Other Pre Specified Outcome: Symptom Burden
Description: Symptom burden was assessed using the PROMIS-29 Sleep Disturbance, Pain Interference, Anxiety, Depression, and Fatigue subscales (0-100) Subscales are averaged into a composite score.The Composite scale ranges from 0 to 100, with higher scores indicating higher symptom burden.
Time Frame: Baseline, Midtreatment, Posttreatment, 3 month follow up, 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group 2 | RESTORE Intervention
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 53.90 (5.23) | 54.90 (5.72)
  Midtreatment | 53.28 (4.99) | 51.63 (6.55)
  Posttreatment | 52.59 (5.69) | 49.42 (7.05)
  3 month follow up | 52.04 (4.65) | 49.04 (6.81)
  6 month follow up | 51.80 (7.32) | 48.11 (7.48)

ADVERSE EVENTS:
Arm/Group | RESTORE Intervention | Control Group 2
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No